CLINICAL TRIAL: NCT04783909
Title: Refractive Outcomes of Phacoemulsification Cataract Surgery in Eyes With Pseudoexfoliation Syndrome
Brief Title: Refractive Outcomes After Cataract Surgery in Eyes With Pseudoexfoliation Syndrome
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Other Study IDs: KE-0254/241/2014
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Refractive Errors; Cataract
Keywords: pseudoexfoliation; phacoemulsification cataract surgery; IOL power calculation formulas
MeSH Terms: conditions — Refractive Errors; Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEX: 42 eyes with PEX syndrome and coexisting cataract
  Interventions: Procedure: Phacoemulsification cataract surgery
- Control: 38 eyes with cataract only
  Interventions: Procedure: Phacoemulsification cataract surgery

INTERVENTIONS:
Procedure: Phacoemulsification cataract surgery — All surgeries were performed using Infinity (Alcon Laboratories, Inc.) under topical anaesthesia by one surgeon through 2.2 mm incision in the upper corneal limbus. The hydroimplantation of IOL to the capsular bag was performed in all cases.

SUMMARY:
To evaluate the refractive outcomes of cataract surgery in PEX syndrome and determine which of the commonly used IOL formulas (SRK/T, Barrett Universal II and Hill-RBF) is the best in predicting postoperative refractive outcomes in PEX.

DETAILED DESCRIPTION:
The primary outcome measure was to compare refractive outcomes (MAE, MedAE, percentage of eyes within certain range of prediction error) in PEX and control eyes. The secondary outcome measure was to determine whether any of IOL power prediction formulas (SRK/T, Barrett Universal II and Hill-RBF) is more precise for these challenging eyes.

ELIGIBILITY:
Inclusion Criteria:

* senile cataract with/without PEX

Exclusion Criteria:

* corneal pathology
* glaucoma,
* corneal astigmatism greater than 2.0 diopters (D),
* previous eye surgery or subjects with decreased vision due to other reasons than cataract (e.g., exudative age-related macular degeneration (AMD), proliferative diabetic retinopathy, inflammatory eye diseases),
* intraoperative complications,
* postoperative corrected distance visual acuity (CDVA) worse than 20/40,
* axial length below 21 mm and above 25 mm,
* dense cataracts or poor fixation requiring ultrasound biometry
* eyes with manifest iridophacodonesis and those in which a capsular tension ring was inserted

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients above 18 yo with senile cataract with/without PEX without coexisting ocular pathologies
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
To compare refractive outcomes in PEX and control eyes. | 3 months
  To measure MAE, MedAE, percentage of eyes within certain range of prediction error after cataract surgery

SECONDARY OUTCOMES:
To determine whether any of IOL power prediction formulas is more precise for these challenging eyes. | 3 months
  To measure the effects of IOL power calculation formulas - SRK/T, Barrett Universal II and Hill-RBF - on postoperative refraction

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Żarnowski, MD, PhD, Professor, Study Chair — Medical University in Lublin

REFERENCES:
- [Derived] Wlaz A, Kustra A, Rozegnal-Madej A, Zarnowski T. Intraocular lens power calculations in eyes with pseudoexfoliation syndrome. Sci Rep. 2021 Sep 24;11(1):19071. doi: 10.1038/s41598-021-98675-5. PMID 34561548